CLINICAL TRIAL: NCT00877136
Title: A Treatment of Unresectable Hepatocellular Carcinoma With TheraSphere®
Status: Completed | Type: Observational
Sponsor: St. Joseph Hospital of Orange (Other)
Responsible Party: Sponsor
Other Study IDs: 08-029 TheraSphere®
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Liver Tumors; Hepatocellular Carcinoma; Hepatoma; Neoplasms
Keywords: Liver tumors; Liver cancer; Adult primary hepatocellular carcinoma; HCC; Hepatoma; Neoplasms
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: TheraSphere® — TheraSphere® consists of insoluble glass microspheres where yttrium-90 is an integral constituent of the glass. TheraSphere® is delivered into the liver tumor through a catheter placed into the hepatic artery. This artery provides the main blood supply to the tumor in the liver. TheraSphere® being unable to traverse the tumor vasculature is embolized within the tumor and exerts a local beta radiation radiotherapeutic effect with relatively limited concurrent injury to surrounding normal tissue.

SUMMARY:
This is an interdisciplinary study that falls into the Humanitarian Use Device category. There are no hypotheses to be tested in this treatment protocol. The study has the following objectives:

1. Provide supervised access to treatment with TheraSphere® to eligible patients with primary cancer to the liver who are not surgical resection candidates.
2. Evaluate patient experience and toxicities associated with TheraSphere® treatment.
3. Measure tumor response rates

DETAILED DESCRIPTION:
The purpose of this protocol is to provide supervised access at this institution to TheraSphere® treatment for a heterogeneous population of patients with unresectable primary liver tumors, with the liver being the only dominant site of disease. Based on experience gained in previous studies and well-established interventional radiology techniques, this protocol allows multiple treatments with TheraSphere® that may be delivered on an inpatient or out patient basis. Patients may receive a single dose to the whole liver, or lobar treatment delivered as a sequence of treatments approximately 30 - 90 days apart. The investigator, working with co-investigators in radiation oncology, interventional radiology and nuclear medicine, will develop a specific treatment plan for each patient, based upon the presenting condition of the patient, the vascular anatomy, and the desired goal of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of hepatocellular carcinoma. The histopathology confirmation criterion may be waived in patients with a radiographically identifiable liver mass with known laboratory or clinical risk factors for cancer or elevated tumor markers such as AFP (clinical diagnosis)
* Surgical evaluation must conclude the patient is not a candidate for resection or ablation.
* ECOG Performance Status Score 0 - 2.
* Age 18 years or older.
* Able to comprehend and provide written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

Any pre-treatment laboratory findings within 15 days of treatment demonstrating:

* Absolute granulocyte count less than or equal to 1,500/ul
* Uncorrected Platelet count less than or equal to 75,000/ul
* Serum creatinine greater than or equal to 3.0 mg/dl
* Serum bilirubin greater than or equal to 2.0 mg/dl
* Any of the following contraindications to angiography and selective visceral catheterization, 1.)History of severe allergy or intolerance to any contrast media, narcotics, sedatives, or atropine, 2.) Bleeding diathesis, not correctable by usual forms of therapy, and/or 3.) Severe peripheral vascular disease that would preclude catheterization.
* Portal hypertension with portal venous shunt away from the liver.
* Evidence of potential delivery of greater than 16.5 mCi (30 Gy absorbed dose) of radiation to the lungs on either: 1) first TheraSphere® administration; or 2) cumulative delivery of radiation to the lungs > 30 Gy over multiple treatments.
* Evidence of any detectable Tc-99m MAA flow to the stomach or duodenum, after application of established angiographic techniques to stop such flow.
* Significant extrahepatic disease representing an imminent life-threatening outcome.
* Severe liver dysfunction (Childs' Classification C) or pulmonary insufficiency (requiring continuous oxygen therapy).
* Active uncontrolled infection
* Significant underlying medical or psychiatric illness.
* Pregnant women may not participate.
* Children may not participate due to lack of clinical experience.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from St. Joseph Hospital of Orange, community members in the St. Joseph Hospital service area and surrounding areas
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2009-02; Primary Completion 2015-02 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Number of patients given access to treatment with TheraSphere. | 24 months
  The number of eligible patients provided with supervised access to treatment with TheraSphere with primary cancer to the liver who are not surgical resection candidates.
Evaluate patient experience with Therasphere. | 24 months
  Evaluation of patient experience and toxicities associated with Therasphere via patient follow-ups with clinician notes.

SECONDARY OUTCOMES:
Tumor response to treatment with TheraSphere® | 24 Months
  Diagnostic imaging studies for assessment of tumor response will be performed according to usual standard of care as established by the referring oncologist.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Wagman, M.D., F.A.C.S., Principal Investigator — St. Joseph Hospital of Orange
Locations (1):
- The Center for Cancer Prevention & Treatment at St. Joseph Hospital of Orange, Orange, California, United States